CLINICAL TRIAL: NCT01939600
Title: Digestibility of Selected Resistant Starches in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Ingredion Incorporated (Industry); University of Toronto (Other); Glycemic Index Laboratories, Inc (Industry); Iowa State University (Other)
Responsible Party: Principal Investigator, Thomas Wolever, Scientist at Keenan Research Centre in the Li Ka Shing Knowledge Institute, Unity Health Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GIL-1322
Record Dates: First submitted 2013-08-29; First posted 2013-09-11 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Malabsorption; Carbohydrate; Ileostomy - Stoma
Keywords: Resistant starch; Ileostomy; In vivo; Carbohydrate digestibility
MeSH Terms: conditions — Malabsorption Syndromes | interventions — high-amylose maize type 2 resistant starch, maize; Amylopectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will undergo all 4 treatments, starch-free breakfast, Hi-Maize 260, Hylon VII and Amioca in randomized order
  Interventions: Other: Starch-free breakfast; Other: Hi-Maize 260; Other: Hylon VII; Other: Amioca

INTERVENTIONS:
Other: Starch-free breakfast — Starch-free breakfast alone
Other: Hi-Maize 260 — Starch-free breakfast plus 55.3g Hi-Maize 260
Other: Hylon VII — Starch-free breakfast plus 56.9g Hylon VII
Other: Amioca — Starch-free breakfast plus 56.4g amioca starch

SUMMARY:
Dietary fiber is a type of carbohydrate which is not digested in the human small intestine. Whole grains are a source of dietary fiber that are used to promote health; however, using whole grains in commercial products results in a different taste and/or texture than the usual products made from refined grains. Thus, other types of high-fiber ingredients have been developed which can be incorporated into food products with less effect on their taste and/or texture. An example of this is resistant starch, defined as starch which is not digested in the human small intestine. The digestibility of starch is usually determined in-vitro; however, there is evidence that such methods may overestimate the amount of resistant starch by as much as 100%. The measurement of the amount of carbohydrate in the ileal effluent, digestive waste, of subjects with an ileostomy is considered to be the best in-vivo method of starch digestibility. The subjects collect ileal effluent during the day during which time they consume a polysaccharide-free diet. There is evidence that resistant starch consumed at breakfast is completely recovered in ileal effluent 8-10hr after consumption. The purpose of this study will be to compare the carbohydrate content recovered in ileal effluent of 10 subjects with a conventional ileostomy.

DETAILED DESCRIPTION:
Dietary fiber consists mainly of carbohydrates which are not digested in the human small intestine. A high intake of dietary fiber is associated with many health benefits including, but not limited to, improved bowel function and reduced risk of weight gain, cardiovascular disease and diabetes. Therefore, there is great interest in the food industry to produce products enriched with dietary fiber to promote health. One way to achieve this is to use more whole grains (wheat, rice, oats, barley) as ingredients in products such as breakfast cereals, breads and food bars. However, the use of whole grains results in products which have a different taste and/or texture than the usual products made from refined grains. Thus, other types of high-fiber ingredients have been developed which can be incorporated into food products with less effect on their taste and/or texture. Examples of such ingredients are inulin (an oligosaccharide containing fructose) and resistant starch. Resistant starch, defined as starch which is not digested in the human small intestine, is present in small amounts (2-5% of total starch) in many normal foods.

Starch is the most abundant energy containing nutrient in the human diet; it consists of 2 types of polysaccharides: amylose, is a linear polymer consisting of long chains of glucose molecules joined by 1-4 linkages; and amylopectin, a highly branched polymer consisting of long chains of glucose molecules joined by 1-4 linkages with numerous 1-6 linkage branch points. Most (70-80%) of the starch in normal starchy foods (eg. cereals and potatoes) is amylopectin. Amylopectin is highly digestible because its branched structure makes it readily able to gelatinize, the process whereby adjacent starch molecules swell and separate from each other under the influence of moist heat (ie. cooking). By contrast amylose is less digestible because its linear structure allows adjacent molecules to associate by hydrogen bonding which reduces their ability to gelatinize. Some types of commercially available resistant starch come from strains of corn which produce starch containing 70 to 100% amylose.

The digestibility of starch is usually determined in-vitro using methods involving digestion of the starch with α-amylase under pH and temperature conditions thought to mimick digestion in the human small intestine. However, there is evidence that such methods may overestimate the amount of resistant starch by as much as 100%. Methods used to estimate starch digestibility in-vivo include the breath hydrogen method and the measurement of the amount of carbohydrate in the ileal effluent of subjects with an ileostomy. The latter is considered to be the best in-vivo method which involves preparation of subjects with a polysaccharide-free diet the day before then consumption of the test carbohydrate with breakfast. Subjects collect ileal effluent during the day during which time they consume a polysaccharide-free diet. There is evidence that resistant starch consumed at breakfast is completely recovered in ileal effluent 8-10hr after consumption. The objective of this study is to determine the amount of carbohydrates in 3 commercially available starches (Hi-Maize® 260, Hylon® VII and Amioca corn starch) which escape digestion in the human small intestine.

ELIGIBILITY:
Inclusion Criteria:

* males or non-pregnant females with a conventional ileostomy
* clinically stable with no clinical evidence of malabsorption

Exclusion Criteria:

* short bowel syndrome
* acute exacerbation of inflammatory bowel disease
* prone to high output with change in diet
* ileostomy created less than 6 months from the first study visit
* subjects using medications which influence gastrointestinal motility or absorption
* any condition which might, in the opinion of Dr. Wolever or Dr. Kim either: 1) make participation dangerous to the subject or to others, or 2) affect the results
* subjects who cannot or will not comply with the experimental procedures
* food allergies of any kind

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Amount of carbohydrate in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Carbohydrate in ileal effluent will be measured using by proximate analysis and expressed in grams.

SECONDARY OUTCOMES:
Amount of fiber in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Fiber is measured using the Englyst method and expressed in grams.
Amount of starch in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Starch will be measured using the Megazyme assay and expressed in grams.

OTHER OUTCOMES:
Amount of fiber in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Fiber will be measured using fiber assay 2009.01 and expressed in grams.
Amount of fiber in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Fiber will be measured using fiber assay 991.43 and expressed in grams.
Amount of starch in ileostomy effluent | Up to 10 hours after starting to consume breakfast
  Starch will be measured by acid hydrolysis and expressed in grams.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Wolever, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada